CLINICAL TRIAL: NCT06353763
Title: Effectiveness of Immersive Virtual Reality Training Versus Traditional Teaching in Pressure Ulcers Care. A Randomized Controlled Pilot Study
Brief Title: Design, Implementation, and Evaluation of Virtual Reality in the Nursing Curriculum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CV
Record Dates: First submitted 2024-03-25; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-01

CONDITIONS: Pressure Ulcer
Keywords: Virtual reality,
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were blinded in their group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention. Virtual reality (Experimental): Immersive virtual reality learning program based on virtual reality glasses
  Interventions: Other: Immersive virtual reality learning program
- Control group: Traditional teaching (No Intervention): Self learning theoretical lesson and traditional teaching with a task trainer, supervised by a teacher.

INTERVENTIONS:
Other: Immersive virtual reality learning program — The immersive virtual reality learning programme was developed by the research team and two nurse experts in chronic wounds, who designed the learning content and script and created six pressure ulcer (PU) cases. Based on the standards of the European Pressure Ulcer Advisory Panel (EPUAP), the National Pressure Ulcer Advisory Panel (NPUAP) and the National Group for the Study and Advice on Pressure Ulcers and Chronic Wounds (GNEAUPP), prevention of healthy skin (case one), management of grade I, II, III and IV PUs (cases two to five) and an infected PU (debridement intervention) were developed. For each case, there was a formative version with immediate feedback and an evaluative one. Before starting the training, the students learned how to use the virtual reality glasses, buttons and joystick by playing a game that trained different dexterity movements. The computer assembly IVR application was developed using Unity 3D and the virtual objects were designed in 3Ds Max.
  Arms: Intervention. Virtual reality

SUMMARY:
The aim of the study is to determine the effectiveness of an immersive virtual reality learning programme for nursing students, based on virtual glasses, in acquiring the competence (knowledge, skills and attitudes) to care for patients with pressure ulcers, and to compare it with the traditional teaching method.

The design was an exploratory randomised controlled trial. The variables used to measure effectiveness were competence and its attributes: knowledge assessment by a multiple-choice test (Pressure Ulcer Knowledge Assessment Tool, Pukat 2.0 instrument), skill performance by direct observation of procedural skills (simulated cases with standardised patients) and satisfaction and usability assessment (Usefulness, Satisfaction and Ease of Use Questionnaire).

DETAILED DESCRIPTION:
The study was a prospective, randomized, double-blind controlled trial conducted from March to May 2022 at a Nursing Faculty. The participants were second-year Nursing Bachelor Degree students from a University in the North of Spain. A convenience sample of students in the second year of the nursing program participated in the study. According to the sample size calculation for a two-tailed independent t-test, conducted using the G*Power 3.1.9 program, with a type I error rate of 0.05, power of 0.80, and an effect size of 0.71, the estimated minimum required sample size was 33. The recommended sample size was 40 participants per group, accounting for a 10% allowance for withdrawals, missing data, and lost follow-up. After registering to enrol in the study, 127 students were screened by the researchers for eligibility. Of these, 99 volunteers met the inclusion criteria and were contacted to schedule the pre-test phase. Following the pre-test assessment, participants were randomly assigned to either the intervention group (50 students) or the control group (49 students) at a 1:1 allocation ratio using a computer-generated assignment. During the study, three participants in the intervention group and two in the control group were excluded due to missing follow-up (refusal to continue in the research), and one student in the control group was removed by statistical analysis. In total, 93 participants were included in the data analysis.

Data was collected from February to May, a period during which the students did not have exams. The demographic information form included fields for age, gender, specific learning related to pressure ulcer care at degree level, and previous experience with virtual reality devices and environments.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in the 2rd year of nursing at the Faculty of Nursing of the University of Navarra and who voluntarily agree to participate in the study.

Exclusion Criteria:

* Students who had acquired the skill of caring pressure ulcers in advance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Knowledge | One month
  The Pressure Ulcer Knowledge Assessment Tool (PUKAT) 2.0 was used to evaluate students' understanding of caring for patients with pressure ulcer problems. The instrument was created and validated by Manderlier (2017). It consists of 25 multiple-choice items, each with a stem containing the problem and five response alternatives. The items are categorized into six relevant themes: 'Aetiology' (6 items), 'Classification and observation' (4 items), 'Risk assessment' (2 items), 'Nutrition' (3 items), 'Prevention of PU' (8 items), and 'Specific patient groups' (2 items). Each correct answer was awarded one point, with a total score of 25. Incorrect answers were not penalised. A higher score indicated a better understanding of PU prevention and care.
Skill performance | One month
  To assess procedural skill in pressure ulcers care, a simulation-based experience (SBE) with a standardized patient was created. The SBE consisted of six cases, each corresponding to one of the six levels of Immersive Virtual Reality (IVR) training, but with different images. Upon entering the classroom, the student had to choose one of six real images, face down, and turn it over to reveal the hazard for the experiment. The simulation-based experience should be completed within ten minutes using the knowledge acquired through self-learning and IVR training. This includes the use of tools such as the Braden scale or the T.I.M.E. (Tissue, infection, moisture, edges) clinical decision support tool to care for the level of pressure ulcers shown in the image. The SBE was evaluated using a 10-item rubric created by the research team and reviewed by a nurse specialist in chronic wounds and pressure ulcers.
Usefulness, Satisfaction, and Ease of Use | One month
  Usability refers to the ease of identifying, comprehending, and using something. To measure the usability and satisfaction of the glasses, we used the Usefulness, Satisfaction, and Ease of Use (USE) questionnaire developed by Lund (2001). The questionnaire assesses four dimensions: usefulness, ease of use, ease of learning, and satisfaction. The USE questionnaire consists of 30 items that assess usability on a 7-point Likert scale ranging from 1 (totally disagree) to 7 (totally agree). The questionnaire has good face validity, reliability, and validity due to its unambiguous and relevant descriptions.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Las Rosas-Salas, Principal Investigator — University of Navarra
Locations (1):
- University of Navarra, Pamplona, Navarre, Spain